CLINICAL TRIAL: NCT04460937
Title: A Phase 1 Trial Combining WEE1 Inhibitor Adavosertib (AZD1775) With Radiation Therapy for Metastatic or Inoperable and Ineligible for Definitive Chemoradiation Esophageal and Gastroesophageal Junction Cancer
Brief Title: Testing the Addition of an Anti-cancer Drug, Adavosertib, to Radiation Therapy for Patients With Incurable Esophageal and Gastroesophageal Junction Cancers
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2020-04698; NCI-2020-04698 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10389 (Other: Ohio State University Comprehensive Cancer Center LAO); 10389 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2020-07-07; First posted 2020-07-08 (Actual); Results first posted 2025-06-08 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-06

CONDITIONS: Clinical Stage III Esophageal Adenocarcinoma AJCC v8; Clinical Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IV Esophageal Adenocarcinoma AJCC v8; Clinical Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVA Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Clinical Stage IVB Esophageal Adenocarcinoma AJCC v8; Clinical Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Clinical Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Distal Esophagus Adenocarcinoma; Gastric Cardia Adenocarcinoma; Metastatic Esophageal Adenocarcinoma; Metastatic Esophageal Squamous Cell Carcinoma; Metastatic Gastroesophageal Junction Adenocarcinoma; Metastatic Malignant Neoplasm in the Brain; Metastatic Malignant Neoplasm in the Leptomeninges; Pathologic Stage III Esophageal Adenocarcinoma AJCC v8; Pathologic Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IIIB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IV Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVA Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Pathologic Stage IVB Esophageal Adenocarcinoma AJCC v8; Pathologic Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Pathologic Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage III Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage III Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IIIB Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IV Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IVA Gastroesophageal Junction Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Esophageal Adenocarcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Esophageal Squamous Cell Carcinoma AJCC v8; Postneoadjuvant Therapy Stage IVB Gastroesophageal Junction Adenocarcinoma AJCC v8; Unresectable Esophageal Adenocarcinoma; Unresectable Esophageal Carcinoma; Unresectable Esophageal Squamous Cell Carcinoma; Unresectable Gastroesophageal Junction Adenocarcinoma
MeSH Terms: conditions — Adenocarcinoma Of Esophagus; Esophageal Squamous Cell Carcinoma; Brain Neoplasms; Meningeal Carcinomatosis | interventions — adavosertib; Radiotherapy; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (radiation therapy, adavosertib) (Experimental): Patients undergo radiation therapy QD 5 days per week for 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive adavosertib PO QD for 2-5 days (depending on dose level) during weeks 1 and 3 of radiation therapy in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Adavosertib; Radiation: Radiation Therapy

INTERVENTIONS:
Drug: Adavosertib — Given PO
  Other Names: AZD 1775; AZD-1775; AZD1775; MK 1775; MK-1775; MK1775
Radiation: Radiation Therapy — Undergo radiation therapy
  Other Names: Cancer Radiotherapy; Energy Type; ENERGY_TYPE; Irradiate; Irradiated; Irradiation; Radiation; Radiation Therapy, NOS; Radiotherapeutics; Radiotherapy; RT; Therapy, Radiation

SUMMARY:
This phase I trial investigates the side effects and best dose of adavosertib and how well it works when given in combination with radiation therapy in treating patients with esophageal or gastroesophageal junction cancer for which no treatment is currently available (incurable). Adavosertib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Radiation therapy uses high energy x-rays to kill tumor cells and shrink tumors. Giving adavosertib together with radiation therapy kill more tumor cells than radiation therapy alone in treating patients with esophageal and gastroesophageal junction cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To identify the maximally tolerated dose of adavosertib (AZD1775) to be used in combination with radiation therapy for patients with esophageal/gastroesophageal junction (GEJ) cancer that is metastatic or inoperable and not eligible for definitive chemoradiation.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity. II. To evaluate the efficacy of AZD1775 when administered in combination with radiation therapy by assessing changes in Ogilvie dysphagia score following treatment, time to second intervention for dysphagia, and overall survival.

III. To identify biomarkers that are predictive for response to experimental therapy.

OUTLINE: This is a dose escalation study of adavosertib.

Patients undergo radiation therapy once daily (QD) 5 days per week for 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive adavosertib orally (PO) QD for 2-5 days (depending on dose level) during weeks 1 and 3 of radiation therapy in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 3 weeks, every 3 months for 2 years, then every 6 months for 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed esophageal cancer (either squamous cell or adenocarcinoma), including Siewert gastroesophageal junction adenocarcinomas types 1 and 2, that is inoperable and not eligible for definitive chemoradiation after multidisciplinary review or have pathologically confirmed or imaging consistent with metastatic disease
* Age >= 18 years. Because no dosing or adverse event data are currently available on the use of AZD1775 in combination with radiation therapy in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1 (Karnofsky >= 70%)
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Hemoglobin >= 9 g/dL
* Platelets >= 100,000/mcL
* Total bilirubin =< 1.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x institutional ULN
* Creatinine =< 1.5 x institutional ULN OR
* Glomerular filtration rate (GFR) >= 60 mL /min/1.73 m^2 unless data exists supporting safe use at lower kidney function values, no lower than 30 mL/min/1.73 m^2
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with new or progressive brain metastases (active brain metastases) or leptomeningeal disease are eligible if the treating physician determines that immediate CNS specific treatment is not required and is unlikely to be required during the first cycle of therapy
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class 2B or better
* Patients able to swallow whole capsules. Patients with esophageal stents and/or feeding tubes are eligible but must be able to swallow whole capsules. Capsules may not be opened or put down a feeding tube
* Patients with a life expectancy > 3 months
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG

  * Resting corrected QTc interval using the Fridericia formula (QTcF) > 480 msec (as calculated per institutional standards) obtained from an ECG (Note: if one ECG demonstrates a QTcF > 480 msec, then a mean QTcF of =< 480 msec obtained from 3 ECGs 2-5 minutes apart, is required at study entry)
  * Patients with congenital long QT syndrome are excluded
* The effects of AZD1775 on the developing human fetus are unknown. For this reason and because other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) for 2 weeks prior to study drug exposure, the duration of study participation, and for 1 month after completing treatment. Women of child-bearing potential must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 1 week of registration. Should a woman become pregnant or suspect she is pregnant while she or her partner is participating in this study, she should inform her treating physician immediately. Men treated or enrolled on this protocol must also agree to use adequate contraception for the duration of study participation and for 3 months after completion of treatment. Male patients should not donate sperm during exposure to study drug and for 3 months after study drug discontinuation
* Ability to understand and the willingness to sign a written informed consent document. Participants with impaired decision-making capacity (IDMC) will also be eligible

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to starting study therapy
* Patients who have not recovered from adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients who are receiving any other investigational agents
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to AZD1775
* Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A4 are ineligible. Because the lists of these agents are constantly changing, it is important to regularly consult a frequently-updated medical reference. As part of the enrollment/informed consent procedures, the patient will be counseled on the risk of interactions with other agents, and what to do if new medications need to be prescribed or if the patient is considering a new over-the-counter medicine or herbal product
* Patients with uncontrolled intercurrent illness
* Patients with psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study because AZD1775 is a WEE1 inhibiting agent with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with AZD1775, breastfeeding should be discontinued if the mother is treated with AZD1775. These potential risks may also apply to other agents used in this study
* Prior thoracic or abdominal radiation therapy for cancer that would result in significant overlap of radiation therapy fields at the discretion of the investigator
* Patients with congenital long QT syndrome or with a history of Torsades de pointes unless all risk factors contributed to Torsades have been corrected. AZD1775 has not been studied in patients with ventricular arrhythmias or recent myocardial infarction
* Eligibility of subjects receiving any medications or substances with the potential to affect the activity or pharmacokinetics of AZD1775 will be determined following review by the principal investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-04-09 (Actual); Primary Completion 2024-03-29 (Actual); Study Completion 2025-12-18 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Eric D Miller, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO
Locations (7):
- United States (7):
  - City of Hope Comprehensive Cancer Center, Duarte, California
  - Northwestern University, Chicago, Illinois
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pittsburgh Cancer Institute (UPCI), Pittsburgh, Pennsylvania
  - University of Utah Sugarhouse Health Center, Salt Lake City, Utah
  - Huntsman Cancer Institute/University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- 150mg Adavosertib, Radiation Therapy; 200mg Adavosertib, Radiation Therapy: Patients undergo radiation therapy QD 5 days per week for 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive adavosertib PO QD for 2-5 days (depending on dose level) during weeks 1 and 3 of radiation therapy in the absence of disease progression or unacceptable toxicity.
  Adavosertib: Given PO
  Radiation Therapy: Undergo radiation therapy
Period: Overall Study
Arm/Group | 150mg Adavosertib, Radiation Therapy | 200mg Adavosertib, Radiation Therapy
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 150mg Adavosertib, Radiation Therapy | 200mg Adavosertib, Radiation Therapy | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 1 | 1 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 2 | 2 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 2 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Planned analysis for the MTD was to employ a BOIN design where the target toxicity rate for the MTD is 25% with 75% dose-elimination cut-off. Due to the study ending early and low enrollment numbers, analysis of MTD was unable to be performed. The data presented is the maximum dose that was reached in the dose-escalation.
Time Frame: After completion of treatment, an average of 3 weeks
Measure: Number; unit: milligrams
Groups:
- All Participants: Patients undergo radiation therapy QD 5 days per week for 3 weeks in the absence of disease progression or unacceptable toxicity. Patients also receive adavosertib PO QD for 2-5 days (depending on dose level) during weeks 1 and 3 of radiation therapy in the absence of disease progression or unacceptable toxicity.
  Adavosertib: Given PO
  Radiation Therapy: Undergo radiation therapy
Arm/Group | All Participants
Number analyzed (Participants) | 4
milligrams | 200

2. Primary Outcome: Number of Adverse Events
Description: Frequency and severity of adverse events and tolerability of the regimen will be collected and summarized with descriptive statistics. The maximum grade for each type of toxicity will be recorded for each patient, and frequency tables will be reviewed to determine toxicity patterns.
Time Frame: From baseline until completion, an average of 6 months
Measure: Number; unit: Number of Events
Arm/Group | 150mg Adavosertib, Radiation Therapy | 200mg Adavosertib, Radiation Therapy
Number analyzed (Participants) | 2 | 2
Number of Events
  Weight loss (Grade 1) | 2 | 3
  Weight loss (Grade 2) | 0 | 1
  Lymphocyte Count Decreased (Grade 1) | 2 | 1
  Lymphocyte Count Decreased (Grade 2) | 1 | 2
  Lymphocyte Count Decreased (Grade 3) | 1 | 2
  Lymphocyte Count Decreased (Grade 4) | 1 | 0
  Trichomonas (Grade 2) | 1 | 0
  Back Pain (Grade 1) | 0 | 1
  Back Pain (Grade 2) | 1 | 1
  Bronchpneumonia (Grade 2) | 1 | 0
  Fatigue (Grade 1) | 1 | 0
  Fatigue (Grade 2) | 1 | 0
  Productive Cough (Grade 1) | 1 | 0
  Productive Cough (Grade 2) | 1 | 1
  Nausea (Grade 1) | 2 | 0
  Nausea (Grade 2) | 1 | 0
  Pericardial Effusion (Grade 2) | 1 | 0
  Increasing Esophageal Pain (Grade 2) | 0 | 1
  Confusion (Grade 1) | 0 | 1
  Confusion (Grade 2) | 0 | 1
  Hyperglycemia (Grade 1) | 1 | 1
  Hyperglycemia (Grade 2) | 0 | 1
  Anorexia (Grade 1) | 1 | 1
  Anorexia (Grade 2) | 0 | 1
  Anemia (Grade 1) | 1 | 1
  Anemia (Grade 2) | 0 | 1
  Hypoalbuminemia (Grade 1) | 3 | 3
  Hypoalbuminemia (Grade 2) | 0 | 1
  Dyspnea (Grade 1) | 1 | 1
  Dyspnea (Grade 2) | 0 | 1
  Sacral Pressure Ulcer (Grade 2) | 0 | 1
  Abdominal Pain (Grade 1) | 1 | 1
  Abdominal Pain (Grade 2) | 0 | 1
  Pneumonitis (Grade 2) | 0 | 1
  Alkaline Phosphate Increased (Grade 1) | 0 | 1
  Alkaline Phosphate Increased (Grade 2) | 0 | 1
  Vomiting (Grade 1) | 3 | 3
  Hypoglycemia (Grade 1) | 1 | 0
  Urinary Urgency (Grade 1) | 1 | 0
  Hematuria (Grade 1) | 1 | 0
  Cough (Grade 1) | 1 | 1
  Alanine Aminotransferase Increased (Grade 1) | 1 | 0
  Bilateral Nipple Pain (Grade 1) | 1 | 0
  Bilateral Breast Pain (Grade 1) | 1 | 0
  Diarrhea (Grade 1) | 1 | 0
  Pain - Right Serratus Anterior Area (Grade 1) | 1 | 0
  Esophagitis (Grade 1) | 1 | 0
  Nasal Congestion (Grade 1) | 1 | 1
  Hypocalcemia (Grade 1) | 0 | 4
  Neck Pain (Grade 1) | 0 | 1
  Dermatitis Radiation (Grade 1) | 0 | 1
  Dizziness (Grade 1) | 0 | 1
  Hypotension (Grade 1) | 0 | 1
  Aspartate Aminotransferase Increased (Grade 1) | 0 | 1
  Blood Lactate Dehydrogenase Increased (Grade 1) | 0 | 1

3. Secondary Outcome: Symptom Relief Rate
Description: Will be calculated with 95% binomial confidence intervals.
Time Frame: After completion of treatment, assessed up to 5 years
Population: Symptom relief data was not measured. Due to low enrollment numbers in phase I and the study not reaching the expansion cohort phase, the study did not collect symptom relief data from participants.
Arm/Group | 150mg Adavosertib, Radiation Therapy | 200mg Adavosertib, Radiation Therapy
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Time to Second Intervention for Dysphagia
Description: Patient dysphagia will be evaluated using the Ogilvie dysphagia score, comparing pre-treatment to post-treatment scores
Time Frame: The time from initiation of therapy to the time of second intervention for dysphagia, assessed up to 5 years
Population: Data was not collected. Data collection was planned for participants in the expansion cohort, and due to the study drug becoming unavailable, the study did not reach the expansion cohort phase. There are no plans for the expansion cohort to be opened at a later date.
Arm/Group | Treatment (Radiation Therapy, Adavosertib)
Number analyzed (Participants) | 0

5. Secondary Outcome: Overall Survival
Description: Overall survival was planned to be analyzed using Kaplan-Meier methods, resulting in median survival times with 95% confidence interval (CI). Due to early termination of the study and low enrollment numbers, planned analysis did not occur. The data presented in this table is the actual months of survival for each participant, measured from enrollment to death.
Time Frame: From date of patient enrollment to death due to any cause, an average of 11.5 months
Measure: Number; unit: months
Arm/Group | Treatment (Radiation Therapy, Adavosertib)
Number analyzed (Participants) | 4
months
  Participant 1 | 28.7
  Participant 2 | 5.07
  Participant 3 | 5.27
  Participant 4 | 8.0

6. Secondary Outcome: Ogilvie Dysphagia Scores
Description: The scores will be summarized and compared using paired t-test or Wilcoxon signed-rank test. Patient dysphagia will be evaluated using the Ogilvie dysphagia score, comparing pre-treatment to post-treatment scores.
Time Frame: At baseline and after completion of treatment
Population: as for outcome 4
Arm/Group | Treatment (Radiation Therapy, Adavosertib)
Number analyzed (Participants) | 0

7. Secondary Outcome: Biomarkers
Description: Will be described graphically or summary measures (e.g. mean and standard errors, or median and range) and compared between responders and non-responders using a two sample t-test or Wilcoxon test if the data is not normally distributed.
Time Frame: Up to 5 years
Population: Biomarkers were not measured. Due to low enrollment numbers in phase I and the study not reaching the expansion cohort phase, the study did not collect biomarker data from participants.
Arm/Group | Treatment (Radiation Therapy, Adavosertib)
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: From study start until completion, an average of 6 months
Arm/Group | 150mg Adavosertib, Radiation Therapy | 200mg Adavosertib, Radiation Therapy
All-Cause Mortality (participants affected / at risk) | 2/2 | 2/2
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 150mg Adavosertib, Radiation Therapy (N=2) | 200mg Adavosertib, Radiation Therapy (N=2)
Weight Loss (Investigations) | 2 (2) | 2 (4)
Vomiting (Gastrointestinal disorders) | 2 (3) | 2 (3)
Nausea (Gastrointestinal disorders) | 2 (3) | 0 (0)
Fatigue (General disorders) | 2 (2) | 0 (0)
Lymphocyte Count Decreased (Investigations) | 2 (5) | 2 (5)
Hyperglycemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hypoglycemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Trichomonas (Infections and infestations) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (2)
Urinary Urgency (Renal and urinary disorders) | 1 (1) | 0 (0)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 2 (2)
Hematuria (Renal and urinary disorders) | 1 (2) | 0 (0)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (3) | 2 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Alanine Aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 1 (1) | 1 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2)
Bilateral Nipple Pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Breast Pain (bilateral) (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Productive Cough (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 1 (1)
Pain - Right Serratus anterior area (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anorexia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Bronchpneumonia (Infections and infestations) | 1 (1) | 0 (0)
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2)
Pericardial Effusion (Cardiac disorders) | 1 (1) | 0 (0)
Hypocalcemia (Metabolism and nutrition disorders) | 0 (0) | 2 (4)
Increasing Esophageal Pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Confusion (Psychiatric disorders) | 0 (0) | 1 (2)
Neck Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Dermatitis Radiation (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Sacral pressure ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Aspartate Aminotransferase Increased (Investigations) | 0 (0) | 1 (1)
Alkaline Phosphate Increased (Investigations) | 0 (0) | 1 (2)
Blood lactate dehydrogenase increased (Investigations) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT04460937/Prot_SAP_000.pdf
  • Informed Consent Form (2022-01-13): https://cdn.clinicaltrials.gov/large-docs/37/NCT04460937/ICF_001.pdf